CLINICAL TRIAL: NCT03692884
Title: Chongqing Diabetes and Its Chronic Complications Registry Study
Brief Title: Chongqing Diabetes Registry Study
Acronym: CDR
Status: Recruiting | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qifu Li, Director of endocrinology, Chongqing Medical University
Other Study IDs: CDR2018
Record Dates: First submitted 2018-07-17; First posted 2018-10-02 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; risk factors; biomarkers; chronic diabetes complications
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Serum, plasma,complete blood cell and urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the risk factors and biomarkers of the microvascular disease，macrovascular disease and neuropathy in patients with diabetes.

DETAILED DESCRIPTION:
This study is a prospective cohort study. About 5000 patients with diabetes from the Chongqing Diabetes Centre,Chongqing,China, will be enrolled for long-term follow-up.Information on socio-demographic parameters, medical history, current drug use,lifestyle factors, anthropometric measurements, metabolic control indicators and diabetes complications examination will be documented. Blood and urine samples will be collected. This study aimed to assess risk factors and biomarkers of occurrence and development of diabetic microvascular disease,macrovascular disease and neuropathy in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of diabetes mellitus（based on the 1999 WHO diagnostic cretirial）;
2. Age younger than 75 years old, gender is not limited;
3. Voluntary to sign on the informed consent.

Exclusion Criteria:

1. pregnant or breast-feeding women;
2. Patients with chronic disease requiring long-term glucocorticoid therapy;
3. Patients with severe infection (except for diabetic foot) or immune dysfunction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects who diagnosed of diabetes mellitus and signed on the informed consent will be enrolled in our study. We intend to enroll hospitalized patients or outpatient with diabetes mellitus from Chongqing Diabetes Centre,Chongqing,China.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
The number of patients whoes Diabetic Kidney disease (DKD) is worsen | 5 years
  Worsen DKD is defined as Urine Albumin Creatinine Ratio （UACR）> 300 mg/g Cr（twice out of three measures）, or 24 hours urinary protein> 300 mg / 24 h, or double serum creatinine level and at least 200μmol/l (2.26 mg/dl), or require renal replacement therapy, or death due to kidney disease.

SECONDARY OUTCOMES:
The number of patients who develop DKD | 5 years
  Diabetic Kidney Disease is defined as UACR > 30 mg/g Cr（twice out of three measures），or estimated Glomerular Filtration Rate（eGFR）<60ml/min/1.73m2.
The number of patients who develop Diabetic Retinopathy | 5 years
  New Diabetic Retinopathy
The number of patients whoes DR is worsen | 5 years
  Worsen DKD is defined as any eye with original Diabetic Rretinopathy aggravated by at least one level, or progress to proliferation retinopathy, or appearance of macular degeneration, or at least one eye with blindness (refer to the WHO standards, the Snellen-chart vision drop to 6/60 or less), or to accept retinal photocoagulation treatment, or accept vitrectomy.
The number of patients who develop Diabetic Neuropathy | 5 years
  Diabetic Peripheral Neuropathy is defined as Neuropathy Symptom Score/Neuropathy Disability Score（NSS/NDS） with at least two positive outcomes, or electromyography examination to identify nerve damage；Diabetic Autonomic Neuropathy is defined as tachycardia at rest (Heart Ratio>100bpm) and postural hypotension (standing position leads systolic blood pressure reduction >20mmHg).
The number of patients who develop Cardiovascular events | 10 years
  Cardiovascular events are difined as death of cardiovascular events, or non-fatal myocardial infarction, or non-fatal stroke, or revascularization procedure (cardiac, carotid, or peripheral), or hospitalization for heart failure.
The number of patients who develop Diabetic foot | 10 years
  Diabetic foot was defined as active diabetic foot problem: ulceration, spreading infection, critical ischaemia, gangrene, suspicion of an acute Charcot arthropathy, or an unexplained hot, red, swollen foot with or without pain.

CONTACTS AND LOCATIONS:
Overall Officials: Qifu Li, phD, Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- Qifu Li, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Lv L, Zhou Y, Chen X, Gong L, Wu J, Luo W, Shen Y, Han S, Hu J, Wang Y, Li Q, Wang Z; Chongqing Diabetes Registry Group. Relationship Between the TyG Index and Diabetic Kidney Disease in Patients with Type-2 Diabetes Mellitus. Diabetes Metab Syndr Obes. 2021 Jul 17;14:3299-3306. doi: 10.2147/DMSO.S318255. eCollection 2021. PMID 34305401